CLINICAL TRIAL: NCT05460234
Title: Non-interventional Study to Collect Real-world Effectiveness, Safety, and Adherence Data on Extended-release Calcifediol (Rayaldee®) in Non-dialysis CKD Patients With Secondary Hyperparathyroidism. Protocol Version 2.0, 06DEC2023
Brief Title: RAYALDEE Non Interventional Study (NIS) on Effectiveness in ND-CKD SHPT Patients
Acronym: PORTRAY
Status: Completed | Type: Observational
Sponsor: Vifor (International) Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Other Study IDs: CS-RAY-2021-0421
Record Dates: First submitted 2022-06-08; First posted 2022-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease
Keywords: hyperparathyroidism; calcifediol
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Cohort: data from medical records up to 3 months prior to ERC treatment start will be retrospectively collected (if available), to provide baseline data and to serve as a basis for evaluating the treatment decision. If relevant baseline data is not available within 3 months preceding treatment start, retrospective documentation can extend to up to 6 months. The observational period of ERC (both retrospective and prospective) is scheduled up to 18 months after treatment start (Protocol v2.0,06Dec2023)

SUMMARY:
The overall study objective is to collect real-world data on the safety and effectiveness of ERC to gradually increase 25D to the level required by Stage 3 and 4 CKD patients.

ERC (Rayaldee), a prolonged-release calcifediol (PRC) formulation, is an orally administered prohormone of active Vitamin D (1,25-dihydroxyvitamin D (1,25D)) designed to increase serum total 25D safely and to a high enough magnitude to reliably reduce elevated PTH in patients with non-dialysis chronic kidney disease (ND-CKD). Clinical studies show that ERC is an effective, well tolerated treatment for secondary hyperparathyroidism (SHPT) in ND-CKD patients with Vitamin D insufficiency or deficiency. ERC gradually raises serum 25D levels, resulting in physiologically regulated increases in serum 1,25D and sustained and progressive reductions in PTH levels, while avoiding clinically meaningful increases in serum phosphate and calcium.

To date, experience with the use of ERC results exclusively from patients from the US and mainly from patients who have participated in clinical trials. It is therefore of major interest to observe the value of ERC in daily use outside of the controlled trial settings in the US as well as in Europe. (Protocol v.2.0,06Dec2023).

DETAILED DESCRIPTION:
Non-interventional, prospective, multicentre, cohort study. Approximately 100 patients diagnosed with ND-CKD with SHPT being treated with ERC according to the SmPC will be included.

The scheduled total study duration is 2.5 years, with a recruitment phase of approximately 1.5 years. The individual prospective observational period per patient is scheduled to last up to 12 months, or up to 18 months for pre-treated patients. The number of observational time points for an individual patient will be dependent on the individual observational period and is assumed to be approximately every 3 months.

A patient is eligible if ERC treatment initiation can coincide with the date of patient inclusion in the study or can happen up to 6 months before patient inclusion in the study. The observational period of ERC treatment will be retrospective if it occurs before study inclusion and prospective for the period after study inclusion. The decision to initiate treatment remains with the treating physician, in line with their normal standard of care, in accordance with the SMPC.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

  * Age ≥18 years
  * Indication for ERC treatment in accordance with the currently approved SmPC.
  * Starting ERC treatment or being on ERC treatment for a maximum of 6 months before inclusion in the study.
  * Stable kidney function in the medical judgment of the investigator

Exclusion Criteria:

Parallel participation in an interventional study

• Enrolment in a prior clinical trial with ERC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enrol patients from approximately 18 sites in Germany. Male or female adult patients with a diagnosis of ND-CKD and SHPT who are due to be treated with ERC according to their physicians usual standard of care and in accordance with the SMPC are eligible.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in 25-hydroxyvitamin D (25D) and iPTH levels | From up to 6 months prior of ERC treatment start to up to 18 months after treatment
  ng/mL or nmol/L, pg/mL or pmol/L
Change in serum calcium level | From up to 6 months prior of ERC treatment start to up to 18 months after treatment
  mg/mL or nmol/L
Change in serum phosphate level | From up to 6 months prior of ERC treatment start to up to 18 months after treatment
  mg/mL or nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Markus Ketteler, Prof., Principal Investigator — Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Locations (16):
- Germany (16):
  - Dialysepraxis Spandau - 01012, Berlin
  - Tagesklinik - Lehrpraxis der Charité Dialyse - Apherese -01007, Berlin
  - Städtisches Klinikum Braunschweig gGmbH -01006, Braunschweig
  - Nierenzentrum Eichstätt MVZ GmbH - 01072, Eichstätt
  - Universitätsklinik Greifswald Klinik und Poliklinik für Innere Medizin A -01066, Greifswald
  - Marien Hospital Herne-Uniklinikum - 01003, Herne
  - MVZ Saarpfalz GmbH - 01008, Homburg
  - Westpfalz-Klinikum GmbH - 01025, Kaiserslautern
  - Nephrologische Gemeinschaftspraxis Baumhackl & Rasche - 01028, Kulmbach
  - Klinikum Landshut -01002, Landshut
  - Universitätsklinikum Mainz - 01004, Mainz
  - Uniklinik Münster, Nephrologische Ambulanz - 01018, Münster
  - Universitätsklinikum Münster, Medizinische Klinik D - 01073, Münster
  - Nephrologisches Zentrum Rendsburg-Eckernförde - 01056, Rendsburg
  - Robert-Bosch-Krankenhaus - 01001, Stuttgart
  - Gim - 01013, Witten

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be requested 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later.
  Data will be indefinitely available for requesting
Access Criteria: A research proposal must be approved by an independent review panel and the study sponsor and researchers must sign a data sharing agreement.

REFERENCES:
- [Background] Petkovich M, Melnick J, White J, Tabash S, Strugnell S, Bishop CW. Modified-release oral calcifediol corrects vitamin D insufficiency with minimal CYP24A1 upregulation. J Steroid Biochem Mol Biol. 2015 Apr;148:283-9. doi: 10.1016/j.jsbmb.2014.11.022. Epub 2014 Nov 22. PMID 25446887
- [Background] Sprague SM, Silva AL, Al-Saghir F, Damle R, Tabash SP, Petkovich M, Messner EJ, White JA, Melnick JZ, Bishop CW. Modified-release calcifediol effectively controls secondary hyperparathyroidism associated with vitamin D insufficiency in chronic kidney disease. Am J Nephrol. 2014;40(6):535-45. doi: 10.1159/000369939. Epub 2015 Jan 7. PMID 25572630
- [Background] Sprague SM, Crawford PW, Melnick JZ, Strugnell SA, Ali S, Mangoo-Karim R, Lee S, Petkovich PM, Bishop CW. Use of Extended-Release Calcifediol to Treat Secondary Hyperparathyroidism in Stages 3 and 4 Chronic Kidney Disease. Am J Nephrol. 2016;44(4):316-325. doi: 10.1159/000450766. Epub 2016 Sep 28. PMID 27676085
- [Background] Sprague SM, Strugnell SA, Bishop CW. Extended-release calcifediol for secondary hyperparathyroidism in stage 3-4 chronic kidney disease. Expert Rev Endocrinol Metab. 2017 Sep;12(5):289-301. doi: 10.1080/17446651.2017.1347501. Epub 2017 Jul 11. PMID 30058895
- [Background] Strugnell SA, Sprague SM, Ashfaq A, Petkovich M, Bishop CW. Rationale for Raising Current Clinical Practice Guideline Target for Serum 25-Hydroxyvitamin D in Chronic Kidney Disease. Am J Nephrol. 2019;49(4):284-293. doi: 10.1159/000499187. Epub 2019 Mar 15. PMID 30878999
- [Background] Cozzolino M, Ketteler M. Evaluating extended-release calcifediol as a treatment option for chronic kidney disease-mineral and bone disorder (CKD-MBD). Expert Opin Pharmacother. 2019 Dec;20(17):2081-2093. doi: 10.1080/14656566.2019.1663826. Epub 2019 Nov 1. PMID 31675257
- [Background] Ketteler M, Ambuhl P. Where are we now? Emerging opportunities and challenges in the management of secondary hyperparathyroidism in patients with non-dialysis chronic kidney disease. J Nephrol. 2021 Oct;34(5):1405-1418. doi: 10.1007/s40620-021-01082-2. Epub 2021 Jun 25. PMID 34170509
- [Background] Cozzolino M, Minghetti P, Navarra P. Extended-release calcifediol in stage 3-4 chronic kidney disease: a new therapy for the treatment of secondary hyperparathyroidism associated with hypovitaminosis D. J Nephrol. 2022 Apr;35(3):863-873. doi: 10.1007/s40620-021-01152-5. Epub 2021 Oct 9. PMID 34626363
- [Background] Fadda G, Germain MJ, Broumand V, Nguyen A, McGarvey N, Gitlin M, Bishop CW, Ashfaq A. Real-World Assessment: Clinical Effectiveness and Safety of Extended-Release Calcifediol. Am J Nephrol. 2021;52(10-11):798-807. doi: 10.1159/000518545. Epub 2021 Oct 27. PMID 34818216